CLINICAL TRIAL: NCT06223607
Title: Dual Antiplatelet Therapy (DAPT) in Patients With Baseline Thrombocytopenia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 036.PHA.2022.D
Record Dates: First submitted 2023-11-13; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Baseline Thrombocytopenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The use of clopidogrel as part of DAPT will be associated with lower bleeding rates compared to ticagrelor in patients with chronic thrombocytopenia requiring Percutaneous intervention (PCI )with Drug Eluting Stent (DES) or Bare Metal Stint(BMS).

DETAILED DESCRIPTION:
Patients with thrombocytopenia are at an increased risk of both bleeding and ischemic events following PCI; however, there is a paucity of data on how to optimally manage these risks. Data indicates that ticagrelor is associated with reduced ischemic outcomes with an accompanying increased risk of bleed in the broader population. This study will assess P2Y12 agent selection in patients with chronic thrombocytopenia to determine if one better balances risks of ischemic and bleeding events following coronary intervention

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* PCI with either DES or BMS during study time period (April 1, 2018 through July 1 2021)
* Thrombocytopenia defined as platelet count <100 x103 /µL on at least one occasion prior to PCI
* At least one dose of DAPT post-PCI with aspirin and either clopidogrel or ticagrelor

Exclusion Criteria:

* Death within 48 hours post-PCI
* DAPT prior to cardiac catheterization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population of 18 years of age ,PCI with either DES or BMS during study time period (April 1, 2018 through July 1 2021) ,Thrombocytopenia on at least one occasion prior to PCI and at least one dose of DAPT post-PCI with aspirin and either clopidogrel or ticagrelor
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2024-08-22 (Estimated); Study Completion 2024-08-22 (Estimated)

PRIMARY OUTCOMES:
Incidence of bleeding | 1 year
  To evaluate the difference in bleeding rates in patients with chronic thrombocytopenia maintained on DAPT with clopidogrel compared to patients maintained on DAPT with ticagrelor.

SECONDARY OUTCOMES:
Incidence of ischemic events | 1 year
  number of ischemic events
All-cause mortality | 1 year
  all-cause mortality in patients with chronic thrombocytopenia maintained on DAPT with clopidogrel compared to patients maintained on DAPT with ticagrelor.
Duration of DAPT | 1 year
  To evaluate the difference in rate of ischemic events and all-cause mortality in patients with chronic thrombocytopenia maintained on DAPT with clopidogrel compared to patients maintained on DAPT with ticagrelor.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Rago Crotty, Pharm D, Principal Investigator — Methodist Midlothian Medical Center
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States